CLINICAL TRIAL: NCT02439853
Title: Communication Bridge Speech Therapy Research Study: Using Internet-Based Speech Therapy to Improve Quality of Life and Access to Care
Brief Title: Communication Bridge Speech Therapy Research Study
Acronym: CB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Alzheimer's Association (Other); The Association for Frontotemporal Degeneration (Unknown); Illinois Department of Public Health (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB23-1336
Record Dates: First submitted 2015-04-23; First posted 2015-05-12 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Progressive Aphasia; Frontotemporal Dementia
Keywords: primary progressive aphasia; progressive nonfluent aphasia; progressive aphasia; frontotemporal dementia; frontotemporal lobar degeneration
MeSH Terms: conditions — Aphasia, Primary Progressive; Frontotemporal Dementia; Primary Progressive Nonfluent Aphasia; Aphasia; Frontotemporal Lobar Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Check-In group (Experimental): Subjects in the Check-In group will undergo three check-in sessions with the speech therapist. These sessions will happen remotely, via video-chat, and will last less than an hour. They will occur at 3-, 4-, and 5-months from the subject's enrollment date.
  Interventions: Behavioral: Monthly Check-in Session
- Control Arm (No Intervention): Subjects in the Control arm will not undergo three check-in sessions with the speech therapist.

INTERVENTIONS:
Behavioral: Monthly Check-in Session — Subjects in the Check-In group will have an online session with a speech-language pathologist 3-, 4-, and 5-months from the subject's enrollment date.
  Arms: Check-In group

SUMMARY:
This is a study on Internet-based video-practice speech and language therapy for persons with primary progressive aphasia (PPA), behavioral-variant frontotemporal dementia (bvFTD), or related conditions.

DETAILED DESCRIPTION:
The purpose of this study is:

1. To evaluate the effectiveness of speech and language therapy on a person's ability to communicate immediately after treatment, 6-months after treatment, and 12-months after treatment.
2. To identify the most effective speech and language therapy strategies for persons with these conditions.
3. To determine the feasibility of Internet-based video-practice of speech and language therapy for persons with these conditions.

The study will involve 12 to 15 session over the course of 12 months. Some of these sessions will be in-person at the Northwestern Cognitive Neurology and Alzheimer's Disease Center (Chicago, IL), while others will take place over the Internet, using an online study portal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia with language as a primary symptom (i.e. aphasia)
* An informant who knows the participant well and can answer questions the participant's communication ability
* Adequate hearing to follow conversation (correction permitted)
* Adequate vision (correction permitted)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-03; Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Functional Communication Abilities | Change from baseline assessment at 2-months, 6-months and 12-months post-treatment
  Functional Communication Abilities will be assessed through questionnaires about the participant's language and communication, neuropsychological testing, and speech and language therapy evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Rogalski, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States